CLINICAL TRIAL: NCT04868578
Title: Efficacy of PyROphosPHate Supplementation to Fight ECtopIc Calcification in PseudoXanthoma Elasticum - PROPHECI-PPI Study
Brief Title: PPI Supplementation to Fight ECtopIc Calcification in PXE
Acronym: PROPHECI-PPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-APN-01
Record Dates: First submitted 2021-03-30; First posted 2021-05-03 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pseudoxanthoma Elasticum
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPI (Experimental): the patient take PPI caps
  Interventions: Dietary Supplement: study treatment PPI
- PPI placebo (Placebo Comparator): The patient take PPI placebo
  Interventions: Dietary Supplement: Placebo comparator

INTERVENTIONS:
Dietary Supplement: study treatment PPI — patient take PPI every day during 12 months
  Arms: PPI
Dietary Supplement: Placebo comparator — patient take PPI placebo every day during 12 months
  Arms: PPI placebo

SUMMARY:
Pseudoxanthoma elasticum (PXE) is a rare inherited metabolic disorder (OMIM 264800, frequency 1/25000) characterized by progressive ectopic calcification of connective tissues. PXE mainly affects the skin (inesthetic papules and plaques in the skin folds), the retina (central blindness), the vasculature (peripheral arterial occlusive disease and stroke) and the renal system (renal lithiasis) in adulthood. Although rarely, early lethal forms have been reported. This chronic and highly disabling condition results from a loss of function of the gene encoding for the ABCC6 membrane transporter primarily expressed in the hepatocytes and renal tubular cells. Recently, it has been reported that PXE was characterized by a 50-60% decrease in the plasma level of inorganic pyrophosphate (PPi), a major physiological anti-calcifying factor. PXE is an incurable disease which therapeutic options are limited to symptomatic treatments to stem the devastating effect of the ectopic calcifications. Recently, encouraging proof of concept studies with animals PXE models and healthy volunteers have shown that, contrary to what was initially reported and thought, the oral administration of PPi salts are able to increase PPi plasma levels, opening up new therapeutic perspectives in PXE. Therefore, we propose to perform the first Phase II randomized controlled trial (RCT) to evaluate the safety and efficacy of a daily and oral administration of PPi salts against placebo in PXE patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years and <65 years), men and women, presenting a clinically and biologically authenticated PXE (genotype + phenotype) according to the international diagnostic criteria (26).
* Efficient contraceptive method in woman of childbearing age at inclusion and during the overall study
* Patient affiliated to a social security insurance
* Signed informed consent
* Patient without acute complication linked or not to the pathology at the time of the study

NON-INCLUSION CRITERIA

* Renal insufficiency (i.e. defined by a renal clearance <30ml / min / 1.73 m²)
* Patients with osteomalacia
* Patients with chronic diarrhea (> 1 month)
* Pregnancy, lactating or fertile women who may wish to become pregnant within three years.
* Any other medical condition that may be considered in the opinion of the Principal Investigator.
* Use of bisphosphonate during last 5 years.
* Hypocalcemia (calcium <2.20 mmol/L and ionized calcium <1.15 mmol/L) *.
* Vitamin D deficiency <35 nmol/L *
* Enrollment in another inteventional clinical trial which could interfere with the present study
* patients (>18 years) protected by law

  * After correcting the hypocalcemia and/or vitamin D deficiency, a participant is again suitable for participation in the trial, as long as the participant meets the inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-12-13 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Arterial calcification score | 12 months
  Using manufacturer dedicated software, the investigator, will determine the calcification score from CT images according to the validated Agatston score method. A threshold of 130 Hounsfield Units for calcium detection will be used for the study. Voxels above this threshold representing arterial wall calcifications will be manually identified and selected by the observer on the CT image. Calcifications mass in the studied arterial segments will be analyzed and quantified. The length and antero-posterior mean diameter of each arterial segment will be determined for further normalization of the calcification score to the arterial wall surface (data expressed as HU/mm2 of arterial surface). The intraclass correlation and Bland-Altman coefficient for inter-observer reliability of the total peripheral artery calcium mass measurement will be determined by scoring 10 random scans by two independent investigators.

SECONDARY OUTCOMES:
clinical observation of dermatological changes | 12 months
  number of patient with dematological changes. Dermatological changes will be monitored by a dermatoscopic study of the skin according to the following protocol: Images will be acquired from commonly affected areas (neck, axilla, antecubital fossae, armpits and periumbilical area) by a contact dermatoscope (SD) with non-polarized light and recorded, as previously described .
  The investigators will ensure that the very same areas are imaged at baseline and at the end of the study. The surface of SD elementary changes featuring yellow papulae (presenting as "dots" or "reticular networks") on digitized images will be compared using an open image processing software (ImageJ, https://imagej.nih.gov/ij/index.html NIH).
clinical observation of ophtalmologic changes | 12 Montths
  Number of patietns with ophtalmologic changes. These changes will be monitored (blinded to treatment) by the occurrence of subretinal neovascularization events, the frequency of anti-VEGF administration and the best-corrected visual acuity (BCVA). A sub-retinal neovascularization event will be defined as any of the following that provide an indication to start or intensify anti-VEGF injections to prevent (further) visual impairment: 1) retinal bleeding suspected to be caused by sub-retinal neovascularization (if needed confirmed by fluorescein angiography); 2) a significant increase in sub retinal or intraretinal fluid; and/or 3) growth of a sub retinal neovascular complex. These events will be scored by the trained ophthalmologist of the PXE reference center (Dr Th Bresson) who will be blinded for the treatment.
vascular changes | 12 months
  Ankle Brachial Index (ABI) at rest: Systolic arterial blood pressure will be recorded using a pneumatic cuff wrapped around the ankle. An ultrasound probe allows recording the blood flow in the left and right ankle arteries (namely posterior and anterior tibial arteries) and brachial arteries supine at rest. The ABI is determined by the ratio between the lowest ankle artery pressure and the highest brachial artery blood pressure.
  A peripheral arterial occlusive disease (PAOD) is defined according to the actual recommendations: an ABI <0.90) and an incompressible arterial wall reflecting mediacalcosis defined by ABI>1.40.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Angers Hospital, Angers
  - Nice Hospital, Nice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clotaire L, Rubera I, Duranton C, Gal J, Chamorey E, Humeau H, Yamani S, Chiaverini C, Willoteaux S, Padovani B, Mourozeau L, Mainguy A, Baillif S, Martin L, Leftheriotis G. The PROPHECI trial: a phase II, double-blind, placebo-controlled, randomized clinical trial for the treatment of pseudoxanthoma elasticum with oral pyrophosphate. Trials. 2025 Jan 29;26(1):30. doi: 10.1186/s13063-024-08666-w. PMID 39881395